CLINICAL TRIAL: NCT01584141
Title: A Multi-Center International Hospital-Based Case-Control Study of Lymphoma in Asia (AsiaLymph)
Brief Title: Study of Lymphoma in Asia
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911206; 11-C-N206
Record Dates: First submitted 2012-04-21; First posted 2012-04-24 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Multiple Myleoma; Lympocytic, Follicular; Leukemia; Hodgkin Lymphoma
Keywords: Leukemia; Lymphoma; Occupational Epidemiology; Molecular Epidemiology; Genetic Polymorphisms
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Leukemia; Hodgkin Disease; Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Asian cases with lymphoid or myeloid neoplasma
- Controls: Controls with selected non-cancer diagnosis who were hospitalized in Hong Kong, Chengdu and Tianjin of Mainland China, and Taiwan

SUMMARY:
Background:

- Lymphoma rates in Asia have been lower than in the West, but rates have been rising in recent years. Most studies of lymphoma patients have been conducted in the West. Less information is available about the factors that might contribute to the rise of lymphoma in Asia. Researchers want to collect medical and personal histories and samples from people who have recently been diagnosed with lymphoma. This information will help them study possible reasons for this increase.

Objectives:

- To collect samples and histories as part of an introductory study of lymphoma in Asia.

Eligibility:

* People between 18 and 79 years of age who have entered study hospitals in Hong Kong, Taiwan, and mainland China for treatment for any type of lymphoma.
* Healthy volunteers between 18 and 79 who have never had lymphoma.

Design:

* Participants will be screened with a physical exam and medical history.
* They will provide blood samples and cheek cell samples for testing.
* Participants will complete a questionnaire about their personal health history. They will answer questions about exposures to chemicals like pesticides. They will also be asked about family medical history and work and residential history. Finally they will answer questions about lifestyle factors like diet and exercise.
* They will give permission for the researchers to see their medical records. Researchers will also have access to any tumor samples collected as part of treatment.

DETAILED DESCRIPTION:
The contribution of environmental, occupational and genetic factors to lymphoma has generated a series of novel findings in studies of Caucasians. However, none of the chemical associations have been conclusively established and the identification of the key, functional alleles in gene regions associated with risk of NHL requires further elucidation. Further, the ability to follow-up, confirm, and extend these observations is limited by the low prevalence and limited range of several important chemical exposures and the high to complete linkage disequilibrium among key candidate genetic loci in Western populations. To optimize the ability to build on and clarify these findings, it is necessary to investigate populations that differ from Caucasians in both exposure patterns and underlying genetic structure. A multidisciplinary case-control study of lymphoma in Asia provides an opportunity to replicate and extend recent and novel observations made in studies among Caucasians in a population that is distinctly different with regard to patterns of key risk factors, including range of exposures, prevalence of exposures, correlations between exposures, and variation in gene regions of particular interest. Thus, a hospital-based case-control study of lymphoma in Eastern Asia (i.e., AsiaLymph) of 4,200 cases and 4,200 controls to be enrolled over a three-year period will be conducted. In addition, 2,000 cases of myeloid leukemias and an additional 2,400 cases with less common lymphoma subtypes will be enrolled as well. The major postulated risk factors for evaluation in this study are chemical exposures (i.e., organochlorines, trichloroethylene, and benzene) and genetic susceptibility. Other factors potentially related to NHL, such as viral infections, UV exposure, medical conditions, and other lifestyle factors will also be explored. A particularly noteworthy aspect of AsiaLymph is central pathology review with immunophenotyping by two of the world s leading lymphoma pathologists, which will enable accurate analysis of findings by molecular and histologic subtypes. AsiaLymph represents the optimal next step in the DCEG lymphoma portfolio. AsiaLymph should confirm and extend previous findings, and yield novel insights into the causes of lymphoma and leukemia in both Asia and the West.

ELIGIBILITY:
* INCLUSION CRITERIA:

Eligible cases will be patients at a participating hospital who are between 18 and 79 years of age at time of initial diagnosis and admitted or treated with incident diagnoses of any lymphoid or myeloid neoplasm including all NHL and Hodgkin disease. Although it is important to understand the etiology of lymphoma in children as well, this undertaking would require additional hospitals, instruments, expertise, and funding that are not currently available to our research team. Adults over the age of 80 are generally among the sickest patients in the hospital and often have multiple comorbidities, which may preclude their participation in an interview of this length. Cases will be permanent residents of the general geographic region that is served by the hospital at the time of diagnosis. Cases will include chronic lymphocytic leukemia/small lymphocytic lymphoma, Waldenstrom macroglobulinemia, plasmacytoma, multiple myeloma, aggressive NK cell leukemia, cutaneous lymphomas, myeloid neoplasms, and immunosuppression-associated cases (such as HIV, post transplant, Methotrexate use).

2,400 lymphoid neoplasm cases will be enrolled with less common subtypes in Asian populations including Hodgkin disease, multiple myeloma, chronic lymphocytic leukemia, and NK/T, T, follicular and marginal zone lymphoma, in order to increase statistical power to study risk factors for these tumors.

EXCLUSION CRITERIA:

Cases with previous diagnosis of lymphoma, such as acute lymphoblastic lymphoma, multiple myeloma, chronic lymphocytic leukemia, and non-Hodgkin lymphoma, are ineligible.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study are Asian cases with lymphoid or myeloid neoplasma and controls with selected non-cancer diagnosis who were hospitalized in Hong Kong, Chengdu and Tianjin of Mainland China, and Taiwan.@@@
Sampling Method: Probability Sample
Enrollment: 13433 (Actual)
Dates: Start 2011-07-05 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of chemical exposures and genetic susceptibility | 2020
  A large-scale evaluation of genes associated with lymphoma in Asian populations that parallels efforts being conducted in Caucasian populations (e.g., currently a genome-wide association study (GWAS)) would be particularly informative because of Asian population genetic differences in patterns of LD and local haplotype structure.
Explore relationship between other factors (viral infections, UV exposure, medical conditions, and lifestyle factors and non-Hodgkin Lymphoma | 2020
  Other factors potentially related to NHL, such as viral infections, UV exposure, medical conditions, and other lifestyle factors will also beexplored.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Lan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- China (2):
  - Tianjin Medical University Cancer Institute & Hospital, Hexi District
  - West China Hospital of Sichuan University, Sichuan
- Queen Mary Hospital, Sai Ying Pun, Hong Kong
- Buddhis Dalin Tzu Chi General Hospital, Dalin Town, Taiwan

REFERENCES:
- [Background] Anderson LA, Pfeiffer R, Warren JL, Landgren O, Gadalla S, Berndt SI, Ricker W, Parsons R, Wheeler W, Engels EA. Hematopoietic malignancies associated with viral and alcoholic hepatitis. Cancer Epidemiol Biomarkers Prev. 2008 Nov;17(11):3069-75. doi: 10.1158/1055-9965.EPI-08-0408. Epub 2008 Oct 28. PMID 18957521
- [Background] Aoki R, Karube K, Sugita Y, Nomura Y, Shimizu K, Kimura Y, Hashikawa K, Suefuji N, Kikuchi M, Ohshima K. Distribution of malignant lymphoma in Japan: analysis of 2260 cases, 2001-2006. Pathol Int. 2008 Mar;58(3):174-82. doi: 10.1111/j.1440-1827.2007.02207.x. PMID 18251781